CLINICAL TRIAL: NCT03327376
Title: Daily Ultrasound-screening for CVC-related Thrombosis in Intensive Care Patients
Brief Title: Daily Ultrasound-screening for CVC-related Thrombosis
Acronym: DUCT
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: z2jzk
Record Dates: First submitted 2017-10-08; First posted 2017-10-31 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2017-10

CONDITIONS: Central Venous Catheter Thrombosis; Critical Illness; Ultrasonography
Keywords: central venous catheters; venous thrombosis; ultrasound; critical care
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Critical Illness; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Characteristic and regularity of CRT: The patients who have a central venous catheterization conduct the daily ultrasound-screening for CVC-related Thrombosis (DUCT).
  Interventions: Device: ultrasound-screening

INTERVENTIONS:
Device: ultrasound-screening — Daily ultrasound-screening for CVC-related thrombosis (DUCT) by compression ultrasound and color doppler ultrasound.

SUMMARY:
The central venous catheters (CVC) related thrombosis is an issue of importance to ICU clinicians.This study conducts the daily ultrasound-screening for CVC-related thrombosis (DUCT).Its aim is to evaluate the characteristic and regularity of the central venous catheters (CVC) related thrombosis in ICU patients, and optimize the screening program of CVC-related thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients at least 18 years of age, expected to need a central venous catheterization for at least 48h in ICU.

Exclusion Criteria:

* Patients with infection or inflammation or local trauma at the insertion site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conduct an observational prospective multicenter study.The patients come from the ICUs of Zhejiang province.
Sampling Method: Probability Sample
Enrollment: 1262 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
the incidence rate of central venous catheters related thrombosis (CRT) | the assessment time will be from the time patients admitted in ICU to the time leaving ICU, less than 6 months.
  the percentage of patients who have CRT in all patients included.

SECONDARY OUTCOMES:
the time when the central venous catheters related thrombosis (CRT) occured | the assessment time will be from the time patients admitted in ICU to the time leaving ICU, less than 6 months.
  which day the CRT is found after central venous catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, MD, Study Director — 2nd Affiliated Hospital, Zhejiang University School of Medicine Institute of Emergency Medicine, Zhejiang University; Weidong Tang, MD, Principal Investigator — The First People's Hospital of Fuyang District; Zhiping Huang, MD, Principal Investigator — Beilun District People's Hospital; Zhaohui Ji, MD, Principal Investigator — The First People's Hospital of Huzhou; Hong Liu, MD, Principal Investigator — Lishui Country People's Hospital; Lingcong Wang, MD, Principal Investigator — The First Affiliated Hospital of Zhejiang University of traditional Chinese Medicine; Mingwei Huang, MD, Principal Investigator — Jinhua Central Hospital; Xingwen Zhang, MD, Principal Investigator — Hunan People's Hospital; Yunchao Shi, MD, Principal Investigator — Affiliated Hospital of Jiaxing University; Renfei Shan, MD, Principal Investigator — Taizhou Hospital; Fuzheng Tao, MD, Principal Investigator — Taizhou Hospital of integrated traditional Chinese and Western Medicine; Yi Wang, MD, Principal Investigator — First People's Hospital of Hangzhou; Qijiang Chen, MD, Principal Investigator — Ninghai First Hospital; Ning Zhang, MD, Principal Investigator — Lishui Country People's Hospital; Jian Hu, MD, Principal Investigator — Pinghu first people's Hospital; Dengpan Lai, MD, Principal Investigator — Affiliated Hospital of Hangzhou Teacher's University; Yingru Lu, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Xudong Zheng, MD, Principal Investigator — The Third Affiliated Hospital of Wenzhou Medical University; Jianbo Gao, MD, Principal Investigator — The First People's Hospital of Fuyang District; Bei Tang, MD, Principal Investigator — Jiande First People's Hospital; Wansheng Li, MD, Principal Investigator — Taizhou Hospital; Xiaoyuan Shen, MD, Principal Investigator — Xiaoshan first people's Hospital; Yukang Song, MD, Principal Investigator — Affiliated Wenling Hospital of Wenzhou Medical University; Guojuan Ding, MD, Principal Investigator — Shaoxing People's Hospital; Feng Wu, MD, Principal Investigator — Zhejiang Quhua Hospital; Xin Tian, MD, Principal Investigator — The Central Hospital of Lishui City; Shaoyi Xu, MD, Principal Investigator — The Second Affiliated Hospital of Jiaxing University; Weijun Fang, MD, Principal Investigator — The Central Hospital of Lishui City; LIfeng Wu, MD, Principal Investigator — Yuyao People's Hospital
Locations (1):
- 2nd Affiliated Hospital, Zhejiang University School of Medicine Institute of Emergency Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faustino EV, Spinella PC, Li S, Pinto MG, Stoltz P, Tala J, Card ME, Northrup V, Baker KE, Goodman TR, Chen L, Silva CT. Incidence and acute complications of asymptomatic central venous catheter-related deep venous thrombosis in critically ill children. J Pediatr. 2013 Feb;162(2):387-91. doi: 10.1016/j.jpeds.2012.06.059. Epub 2012 Aug 9. PMID 22883418
- [Background] Lee AY, Kamphuisen PW. Epidemiology and prevention of catheter-related thrombosis in patients with cancer. J Thromb Haemost. 2012 Aug;10(8):1491-9. doi: 10.1111/j.1538-7836.2012.04817.x. PMID 22703114
- [Background] Refaei M, Fernandes B, Brandwein J, Goodyear MD, Pokhrel A, Wu C. Incidence of catheter-related thrombosis in acute leukemia patients: a comparative, retrospective study of the safety of peripherally inserted vs. centrally inserted central venous catheters. Ann Hematol. 2016 Dec;95(12):2057-2064. doi: 10.1007/s00277-016-2798-4. Epub 2016 Aug 20. PMID 27542955
- [Result] Parienti JJ, Mongardon N, Megarbane B, Mira JP, Kalfon P, Gros A, Marque S, Thuong M, Pottier V, Ramakers M, Savary B, Seguin A, Valette X, Terzi N, Sauneuf B, Cattoir V, Mermel LA, du Cheyron D; 3SITES Study Group. Intravascular Complications of Central Venous Catheterization by Insertion Site. N Engl J Med. 2015 Sep 24;373(13):1220-9. doi: 10.1056/NEJMoa1500964. PMID 26398070
- [Result] Gentile A, Petit L, Masson F, Cottenceau V, Bertrand-Barat J, Freyburger G, Pinaquy C, Leger A, Cochard JF, Sztark F. Subclavian central venous catheter-related thrombosis in trauma patients: incidence, risk factors and influence of polyurethane type. Crit Care. 2013 May 29;17(3):R103. doi: 10.1186/cc12748. PMID 23718723